CLINICAL TRIAL: NCT06850012
Title: The Effects of an Education Program Based on Meleis's Transition Theory on Perceived Stress, Professional Self-Efficacy, and Social Adaptation of Migrant Turkish Nurses in Germany
Brief Title: Meleis-Based Training: Perceived Stress, Professional Self-Efficacy, and Social Adaptation of Migrant Turkish Nurses
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Buse Karabulut, PhD Candidate, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 30.01.2025/046
Record Dates: First submitted 2025-02-23; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Mmigrant Nurses' Adaptation and Perceived Stress; Transition Theory in Immigrant Nurses; Social Adaptation and Stress in Immigrant Nurses; Professional Self-Efficacy
Keywords: Transition Theory; Immigrant Nurses; Perceived Stress; Professional Self-Efficacy; Social Integration
MeSH Terms: conditions — Social Adjustment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This study is an open-label trial, meaning that participants, care providers, and investigators are aware of group assignments. However, the data analysis will be conducted by an independent statistician who will be blinded to group allocation to ensure an unbiased assessment of the study outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Meleis' Transition Theory-Based Educational Program (Experimental): This arm will receive a 7-week online educational program based on Meleis' Transition Theory. The program is designed to support immigrant nurses in adjusting to the challenges associated with migration, enhancing social integration, managing stress, and improving professional self-efficacy. The intervention will be conducted entirely online, with participants split into three groups (12-12-11 participants per group). Each weekly session will last approximately 45-50 minutes and will include interactive activities such as group discussions, case studies, and short practical exercises, including breathing exercises to encourage active participation.
  The goal of this program is to provide participants with the tools and strategies to navigate the transition into their new professional and personal environment, improve their stress management, and foster a greater sense of professional self-efficacy and social belonging.
  Interventions: Behavioral: Meleis' Transition Theory-Based Educational Program
- Control Group (No Intervention): this group will not participate in the educational program. Participants will be assessed based on their current status, with factors such as immigrant perception, stress levels, and social integration being observed. The effect of factors other than the education program on these variables will be evaluated.

INTERVENTIONS:
Behavioral: Meleis' Transition Theory-Based Educational Program — This intervention is a 7-week online educational program based on Meleis' Transition Theory, aimed at helping immigrant nurses understand and cope with migration challenges, improve social integration, manage stress, and enhance professional self-efficacy. The program will be divided into three groups (12-12-11 participants), and it will include interactive sessions, group discussions, and practical activities such as breathing exercises to promote active participation and engagement.
  Arms: Meleis' Transition Theory-Based Educational Program

SUMMARY:
This study aims to evaluate the effects of an education program based on Meleis's Transition Theory on perceived stress, professional self-efficacy, and social adaptation among migrant Turkish nurses in Germany. The program will provide training and support to help these nurses manage the challenges of adapting to a new professional and social environment. Participants will engage in a series of educational sessions designed to enhance their coping skills, improve their professional confidence, and reduce perceived stress. The results of the study will contribute to the development of strategies to enhance social adaptation in nursing practice, improve healthcare quality, and support the professional development and migration adaptation processes of migrant nurses. This is a randomized controlled experimental study that examines the effects of an education program based on Meleis's Transition Theory on perceived stress, professional self-efficacy, and social adaptation of Turkish migrant nurses who have migrated to Germany to work.

DETAILED DESCRIPTION:
AIM AND SIGNIFICANCE OF THE PROJECT:

To address the shortage of skilled labor, the German government passed a law in 2020 (Fachkräfteeinwanderungsgesetz) regarding the immigration of skilled workers from outside the European Union to Germany (Bundesregierung der Bundesrepublik Deutschland, 2019). This law facilitates the immigration of nurses and other skilled workers, and currently, Germany and the United Kingdom are among the countries with the highest number of migrant nurses (OECD, 2016). As of 2023, migrant nurses constitute 14.5% of the nursing workforce in Germany, with Turkish nurses playing a significant role in this group (Bibliomed Pflege, 2023).

Migrant nurses face a series of transition processes such as international migration, learning a new language, adapting to a different culture, and adjusting to a new healthcare system and work environment. These processes involve not only individual transformation but also serious challenges in professional life and social integration (Nortvedt et al., 2020; Schilgen et al., 2019; Villamin et al., 2024; WHO, 2020). Issues such as language barriers, lack of social support, discrimination, inadequate orientation processes, and excessive workloads complicate the integration of migrant nurses (Davda et al., 2018; Smith et al., 2022).

These challenges have negative effects not only on psychological well-being but also on professional satisfaction and perceptions of competence. For example, differences in educational levels and insufficient language skills can lead to a loss of professional skills, feelings of devaluation, and general dissatisfaction among nurses (Davda et al., 2018). Additionally, changes in living conditions and difficulties adjusting to climate conditions further complicate the overall adaptation processes for migrant nurses (Villamin et al., 2024). It is believed that these factors may increase the perceived stress levels among migrant nurses, leading to deficiencies in social adaptation and perceptions of professional competence. In this context, the process of adapting to perceived differences is considered a complex transition process that should be addressed not only through personal efforts but also through supportive strategies. Meleis's Transition Theory provides a framework for understanding the effects of major life changes - i.e., transition processes - on health and well-being (Meleis, 2010).

This study aims to explore the transition processes of migrant nurses in Germany using Meleis's Transition Theory, focusing on factors such as stress, adaptation, and self-efficacy, to gain a deeper understanding of how to support them during these transitions. The results of this study will contribute to the development of strategies to enhance social adaptation in nursing practice, improve healthcare quality, and support the professional development and migration adaptation processes of migrant nurses. This is a randomized controlled experimental study that examines the effects of an education program based on Meleis's Transition Theory on perceived stress, professional self-efficacy, and social adaptation among Turkish migrant nurses who have migrated to Germany for work.

GENERAL INFORMATION:

As the global shortage of nurses grows, the World Health Organization (WHO) predicts that by 2035, the global demand for nurses will reach 12.9 million. Nurses migrate for various reasons (financial, professional, political, social, and personal) (Dywili et al., 2013). Today, one in every eight nurses works outside their country of birth or education (WHO, 2020). These nurses are referred to in the literature as internationally educated nurses, foreign nurses, or migrant nurses (Dywili et al., 2013; Villamin et al., 2024; WHO, 2020).

Nurse migration has both positive and negative impacts on individuals and healthcare systems (Li et al., 2014). Migrant nurses can facilitate the transfer of knowledge and skills between source and destination countries, contribute to the labor market, and enrich healthcare services through cultural diversity. Nurses who typically migrate to developed or developing countries for better job, income, and education opportunities are driven by factors such as career prospects, cultural diversity, and economic contributions (Agbede & Asmah, 2024; Li et al., 2014; Villamin et al., 2024). However, alongside these positive aspects, they encounter numerous challenges during their integration process in the destination country and require support (Agbede & Asmah, 2024). For example, when financial incentives lead to economic recovery, or when partially achieved, other needs such as family welfare, community support, recreation, and professional satisfaction may become more important (Villamin et al., 2024). Migrant nurses face challenges such as adaptation difficulties, language barriers (Nortvedt et al., 2020; Schilgen et al., 2019), lack of social support, discrimination (Davda et al., 2018; Smith et al., 2022; Villamin et al., 2024), insufficient orientation processes, excessive workload, harsh living conditions, and difficulties adapting to climate (Villamin et al., 2024). Additionally, differences in educational levels, language skills, and cultural disparities are known to lead to dissatisfaction, devaluation, and loss of professional skills (Davda et al., 2018).

A study conducted with Filipino migrant nurses reported that nurses felt devalued in the countries they migrated to and struggled with language learning and finding housing or work (Nortvedt et al., 2020). Results from a study on migrant nurses in Germany found that language differences were identified as a major stress factor affecting teamwork and nurse-patient relationships (Schilgen et al., 2019). Furthermore, in Germany, differences in work environments, professional competence, ethical understanding, language barriers, cultural alienation, high perceived pressure for adaptation, and changes in professional identity are also issues that can accompany the process (Lauxen et al., 2019). In summary, migrant nurses face challenges related to adapting to a new culture and work environment, and they deal with numerous stress factors during this process. The challenges faced by migrant nurses not only affect their interactions with colleagues and patients but also their cultural adaptation and job satisfaction. Therefore, it is essential to implement and evaluate strategies that support the integration and well-being of migrant nurses (Al-Btoush & El-Bcheraoui, 2024).

Transition, in the literature, is defined as the process of an individual moving from one state or status to another, including the time span, phases, and how the individual perceives this process. In this context, the migration of nurses to practice in a different country is a transition process (Meleis, 2010). Migrant nurses undergo various transition processes, such as international migration, living with a new language, adapting to a new culture, adjusting to a new healthcare system, and integrating socially (WHO, 2020). These transitions are long-term processes that require adaptation to new roles and situations. An individual's transition may be influenced positively or negatively by others, and the support needs of each individual during the transition process differ (Meleis, 2019).

Nurses are at the heart of change and transition processes. They are representatives of a profession that supports individuals who encounter change and those preparing for it (Meleis, 2010, 2019). Immigrant nurses become individuals who need support to successfully adapt to a new culture, different working conditions, and professional environments in this process. This highlights the importance of professional solidarity as well as strategies, resources, and knowledge sharing to support the adaptation of immigrant nurses (Dywili et al., 2013; Villamin et al., 2024; WHO, 2020).

In light of this information, Meleis' Transition Theory can provide a framework to understand the perceived stress, professional self-efficacy, and social adaptation, which are critical dimensions in the professional transition processes of Turkish nurses who have migrated to Germany. It can also evaluate and support the difficulties they experience in these processes. Most studies on immigrant nurses in the international literature are qualitative (Ryan, 2008; Schilgen et al., 2019), reviews (Al-Btoush & El-Bcheraoui, 2024; Correa-Betancour et al., 2024; Smith et al., 2022), or case reports (Lauxen et al., 2019), and recent studies show limitations in their quantitative nature (Al-Btoush & El-Bcheraoui, 2024; Correa-Betancour et al., 2024; Lauxen et al., 2019; Schilgen et al., 2019; Smith et al., 2022). In the national literature, no studies focusing on immigrant nurses have been found.

Considering that a large part of the existing literature consists of qualitative, review, or case report studies, and there is no study focusing on this issue in the national context, it is important to note that nurses, who become individuals in need of support due to challenges such as language barriers, different professional standards, social isolation, and cultural differences after migration. Thus, investigating the effects of a training program designed within the framework of Meleis' Transition Theory on perceived stress, professional self-efficacy, and social adaptation through a randomized controlled experimental design constitutes the unique aspect of this study.

METHOD OF THE THESIS:

1. Research Type The research is planned to be conducted as a randomized controlled experimental study to determine the effects of an educational program developed within the framework of Meleis's Transition Theory on perceived stress, professional self-efficacy, and social adaptation of Turkish nurses who have immigrated to Germany to work.
2. Research Hypotheses H₀₁: The educational program developed within the framework of Meleis's Transition Theory does not affect the perceived stress levels of Turkish immigrant nurses.

   H₁₁: The educational program developed within the framework of Meleis's Transition Theory affects the perceived stress levels of Turkish immigrant nurses.

   H₀₂: The educational program developed within the framework of Meleis's Transition Theory does not affect the professional self-efficacy levels of Turkish immigrant nurses.

   H₁₂: The educational program developed within the framework of Meleis's Transition Theory affects the professional self-efficacy levels of Turkish immigrant nurses.

   H₀₃: The educational program developed within the framework of Meleis's Transition Theory does not affect the social adaptation levels of Turkish immigrant nurses.

   H₁₃: The educational program developed within the framework of Meleis's Transition Theory affects the social adaptation levels of Turkish immigrant nurses.
3. Research Variables Dependent variables: perceived stress, professional self-efficacy, and social adaptation levels.

   Independent variable: the educational program implemented within the framework of Meleis's Transition Theory.
4. Research Location and Characteristics There are various application methods for nurses who have immigrated to Germany. One of these is the individual application process for equivalence procedures. In this process, nurses can apply to practice their profession in Germany by collecting necessary documents and meeting requirements such as language proficiency. Alternatively, immigrant nurses can receive support from equivalence agencies to manage the application process. One of these centers is the Sprachportal Akademie, located in Wetzlar. The research will be conducted at the Sprachportal Akademie Wetzlar, located in Germany, on Turkish immigrant nurses residing in Gießen.
5. Population and Sample The population of the research will consist of Turkish immigrant nurses who have immigrated to Germany and are served by Sprachportal Akademie, providing consultancy services and language courses, and who have immigrated 3 to 24 months ago. The reason for excluding the first three months is that this period is known as the "crisis period," during which challenges such as language barriers, culture shock, social isolation, and adaptation to work and living conditions are most intense. Therefore, excluding individuals in this period is preferred to avoid the influence of early-stage crisis effects on the results. The two-year upper limit is determined based on the idea that the adaptation process stabilizes after this time and individuals have largely integrated into their post-migration lives (Oberg, 1960).

   Due to the limited number of studies conducted on immigrant nurses, the sample size was determined by considering the participant number in Meleis's studies, which usually involved similar sample sizes (typically around 30 participants). Considering potential dropouts, 10% additional participants will be included in each group, leading to a total of 70 participants: 35 in the intervention group (divided into 3 subgroups) and 35 in the control group. After data collection, a post-hoc power analysis will be conducted to assess the actual power level of the study and effect size. This analysis will aim to further confirm the statistical sufficiency and reliability of the findings.

   Inclusion Criteria:
   * Voluntarily agreeing to participate.
   * Aged 18 and over.
   * Immigrated to Germany as a nurse.

   Exclusion Criteria:
   * Diagnosed with a mental disorder that would impede participation.
   * Refusing to participate in the research.

   Termination Criteria:
   * Voluntarily withdrawing from the research or sessions.
   * Failing to attend 2 or more sessions or discontinuing the program.
   * Failing to complete the measurement tools, leaving them incomplete.

   Randomization:

   In this research, randomization for assigning participants to intervention and control groups will be conducted using a completely random system, carried out by a person independent of the research. Participants will be given unique numbers, which will then be randomly assigned to the groups using an online program (e.g., http://www.randomizer.org). This method ensures that participants are randomly placed in groups, increasing the objectivity of the study and minimizing initial differences between the groups.
6. Data Collection Tools Data will be collected using a Personal Information Form, the Perceived Stress Scale-10, the Nursing Professional Self-Efficacy Scale, and the Social Adaptation Scale for Immigrants. Preliminary applications of the data collection and intervention tools will be conducted with 2 immigrant nurses, and final adjustments will be made to the data collection tools.

   Personal Information Form:

   The Personal Information Form was developed by the researcher based on the literature (Agbede & Asmah, 2024; Jepsen et al., 2024) and aims to assess the basic demographic characteristics, language proficiency, social adaptation level, and general stress levels of Turkish nurses who have immigrated to Germany. The form consists of 14 questions, including age, gender, marital status, education level, length of residence in Germany, reasons for immigration, German language proficiency, self-perceived German speaking ability, social adaptation, professional competence perceptions, general stress levels, and daily life stress sources.

   Perceived Stress Scale-10:

   Developed by Cohen, Kamarck, and Mermelstein (1983), the Perceived Stress Scale (PSS) is designed to measure how stressful individuals perceive situations in their life. Responses range from "Never (0)" to "Very often (4)". The scale includes 10 items, with 7 positively phrased items scored in reverse. The maximum score on the PSS-10 is 40, and the minimum is 0. Higher scores indicate higher perceived stress. The Turkish adaptation of the PSS-10 has demonstrated high reliability and validity (Eskin et al., 2013).

   Nursing Professional Self-Efficacy Scale:

   Developed by Caruso et al. (2016), the Nursing Professional Self-Efficacy Scale (NPSES) consists of two subdimensions and 19 items. Responses range from "Strongly disagree (1)" to "Strongly agree (5)". The subdimensions are Quality of Care (e.g., Items 1, 3, 4, 5, etc.) and Professional Situations (e.g., Items 2, 10, 11, etc.). A higher score indicates a higher perception of professional self-efficacy. The Turkish adaptation showed good reliability and validity, with a Cronbach's Alpha coefficient of 0.87 (Vicdan Kacaroğlu & Taştekin, 2019).

   Social Adaptation Scale for Immigrants:

   Developed by Kaya (2022), this scale measures the social adaptation levels of immigrants with 28 items. It assesses various psychological, social, and individual factors immigrants face in their adaptation process. The scale uses a 5-point Likert scale, with items reversed in scoring for certain factors. Higher scores indicate better social adaptation.
7. Data Collection

   Data will be collected between June 2025 and June 2026. The scales (Personal Information Form, Perceived Stress Scale-10, Nursing Professional Self-Efficacy Scale, and Social Adaptation Scale for Immigrants) will be administered as a pre-test to both the intervention and control groups. After the initial measurements, the intervention phase will proceed as follows:
   1. Intervention Group: Participants will be assigned randomly, and the intervention group will be further divided into three subgroups. Each subgroup will undergo a 7-week online educational program consisting of 45-60 minute weekly sessions. The content will cover topics such as immigration and social adaptation, cultural awareness, stress management, professional self-efficacy, and social support. The program will include PowerPoint presentations, exercises, discussions, and experience-sharing. A WhatsApp group will be created to facilitate communication and information exchange during the program. Pre- and post-tests will be conducted using the same measurement tools.
   2. II. Interventions for the Control Group The control group will undergo the same initial measurements as the intervention group, which includes the Personal Information Form, the Perceived Stress Scale-10, the Nursing Professional Self-Efficacy Scale, and the Social Adaptation Scale for Immigrants. A WhatsApp group will be created for the control group for informational purposes, but no education or intervention will be provided through the group. Participants will be able to contact the researcher individually for any necessary support. Apart from this, no interventions will be made with the control group during the 7-week period. After the intervention group completes their training, the control group will also complete the final measurement, which includes the Perceived Stress Scale-10, the Nursing Professional Self-Efficacy Scale, and the Social Adaptation Scale for Immigrants. Following the educational program, the control group will be provided with the educational materials, and if needed, the program will be implemented for them.
8. Preliminary Application In order to assess the appropriateness of the data collection tools and the effects of the Meleis's Transition Theory-based educational program on participants, a preliminary application will be conducted with two participants from each group. This preliminary application will be carried out before the 7-week training process to identify any issues with the program's content or methodology. If any changes need to be made during the preliminary application, such as difficulties or deficiencies related to data collection, educational materials, or methods, the materials and content will be reviewed and updated accordingly. If participants provide feedback on the duration or frequency of the training, the session durations will be adjusted.
9. Data Analysis The data obtained in the study will be analyzed using computer-based methods. Normal distribution assumptions will be considered when applying hypothesis tests. The normality of the data will be evaluated using the Shapiro-Wilk test. Descriptive statistical methods (mean, standard deviation, frequency) will be used when evaluating the study data. When the data is normally distributed, the Independent Samples t-Test will be used for comparisons between two groups, and Repeated Measures Analysis of Variance (ANOVA) will be used for analyzing repeated measurements. Pearson Correlation Analysis will be applied to evaluate relationships between continuous variables. If the data does not show normal distribution, the Mann-Whitney U Test will be used for comparing quantitative data between two groups, and the Friedman Test will be applied for repeated measurements. Spearman Correlation Analysis will be used to assess relationships between continuous variables. A significance level of p<0.05 will be considered.
10. Ethical Aspects of the Research Ethical approval for this study was obtained from the Erciyes University Social and Humanities Ethics Committee (Document no-046). Institutional permission was granted by Sprachportal Akademie. Informed verbal and written consent will be obtained from individuals voluntarily participating in the study. It will be clearly stated that individuals who refuse to participate or wish to discontinue at any stage may withdraw from the study.

During the research process, participants in both the intervention and control groups will be able to continue their regular routines. At the end of the study, educational materials will also be provided to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Participants who voluntarily agree to participate in the study. Aged 18 years or older. Immigrants who have migrated to Germany as nurses.

Exclusion Criteria:

* Individuals with a mental health disorder that could prevent participation in the study.

Those who do not consent to participate in the study.

Termination Criteria:

Participants who voluntarily withdraw from the study or sessions. Participants who miss two or more sessions or discontinue the program. Participants who do not complete the measurement tools or leave them incomplete.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Social Integration (using the Social Integration Scale for Immigrants) | From the start of the educational program to the end of the 7-week intervention period
  This scale measures the level of social integration and community involvement of immigrant nurses. The study will assess whether the educational program has a positive effect on participants' social integration.

SECONDARY OUTCOMES:
Perceived Stress | From the start of the educational program to the end of the 7-week intervention period
  his scale measures the level of stress perceived by immigrant nurses in their daily lives. The study will monitor whether the educational program results in a change in participants' stress levels.
Nursing Professional Self-Efficacy | From the start of the educational program to the end of the 7-week intervention period
  Nursing Professional Self-Efficacy Scale measures the participants' perceived ability to perform nursing tasks. The study will investigate whether the educational program influences participants' professional self-efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Sprachportal Wetzlar, Wetzlar, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared after study completion, upon request, in compliance with ethical guidelines and confidentiality agreements. The shared data will be anonymized and made available for research purposes through a data repository or similar platform. The IPD will not include any personally identifiable information (PII) to ensure participant privacy.
Supporting Information: Study Protocol, SAP, CSR